CLINICAL TRIAL: NCT03681080
Title: Understanding Impaired Concentration, Attentional Deficits and Their Pathophysiology in Postural Orthostatic Tachycardia Syndrome (POTS) and Other Autonomic Neuropathies (POTSKog-Study Aachen)
Brief Title: Concentration and Attentional Deficits in POTS and Other Autonomic Neuropathies
Acronym: POTSKog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Andrea Maier, Dr. Andrea Maier, Principal Investigator, RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-006
Record Dates: First submitted 2018-09-10; First posted 2018-09-21 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Autonomic Failure; Dysautonomia; Cognitive Impairment; Ehlers-Danlos Syndrome; Postural Tachycardia Syndrome; Pure Autonomic Failure
MeSH Terms: conditions — Pure Autonomic Failure; Autonomic Nervous System Diseases; Cognitive Dysfunction; Ehlers-Danlos Syndrome; Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lying (No Intervention): cognitive tests are performed during lying in all groups (SFN, AAN, EDS, POTS and controls)
- standing (No Intervention): cognitive tests are performed during active Standing in all groups (SFN, AAN, EDS, POTS and controls)
- crossed legs (Experimental): cognitive tests are performed during leg crossing in all groups (SFN, AAN, EDS, POTS and controls)
  Interventions: Procedure: leg crossing

INTERVENTIONS:
Procedure: leg crossing — As Counter maneuvre legs will be crossed and cognitive tests will be performed.
  Arms: crossed legs

SUMMARY:
People with POTS, autoimmune autonomic neuropathy (AAN), pure autonomic failure (PAF), SFN and Ehlers Danlos Syndrome (EDS) do not only suffer from orthostatic symptoms such as dizziness, headache, neck pain, blurred vision or (pre-) syncope. They also experience deficits in attention and concentration (more precisely deficits in selective perspective, operating speed, executive functions and memory performance) mainly in upright position. Only few studies concerning cognitive impairment in autonomic neuropathies, their frequency, aetiology and therapy exist. Many patients concerned, especially with POTS, report attention deficits and "brain fog" with problems in their everyday life and work, predominantly in upright posture. Specific symptomatic or medical therapies do not exist. Medical treatment with Modafinil is discussed and part of a current study at Vanderbilt Autonomic Dysfunction Centre (1-5). The investigators want to investigate if problems of concentration, attention and/or cognitive dysfunction exist in people with POTS, AAN, SFN and EDS compared to healthy controls (HC). Thus the investigators use detailed clinical, autonomic and neuropsychological tests in different body positions (lying, sitting and standing) as also acute therapy (leg crossing).

DETAILED DESCRIPTION:
We are still recruting healthy controls and patients with autoimmune autonomic neuropathy in order to perform titl table examination and laboratory testing on day one, ono an empty stomach, without morning medication. Cognitive testing is performed on day two after randomization in three groups: lying, standing and standing with legs crossed.

ELIGIBILITY:
Inclusion Criteria:

* AAN, SFN, hEDS, POTS or healthy control
* diagnosis in our clinic on the basis of anamnesis, clinical data as neurological examination, tilt table, QST, skin biopsy, norepinephrine values, vitamine B12, antibodies

Exclusion Criteria:

for all participants

* pregnancy, nonage,severe heart insufficiency, deep brain Stimulation, pace maker, drug consumption, large fibre polyneuropathy for controls
* medication influencing blood pressure, psychiatric disease, synkopes or dizziness, neurological disorders esp. polyneuropathy, dementia, vitamine or iron deficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
cognitive function: Stroop, TMT A und B | during intervention (Leg crossing)
  Change of results of cognitive function tests lying compared to standing and leg crossing

SECONDARY OUTCOMES:
blood pressure Change (mmHg) | during intervention (Leg crossing)
  Change between blood pressure lying compared to compared to standing and leg crossing
Heart frequency Change (B/min) | during intervention (Leg crossing)
  Change between heart frequency lying compared to compared to standing and leg crossing
cerebral blood flow velocity | during intervention (Leg crossing)
  Change between cerebral blood flow compared to compared to standing and leg crossing

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Maier, Dr., Principal Investigator — Universitiy hospital RWTH Aachen, Department of Neurology
Locations (1):
- University Hospital, RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart JM, Del Pozzi AT, Pandey A, Messer ZR, Terilli C, Medow MS. Oscillatory cerebral blood flow is associated with impaired neurocognition and functional hyperemia in postural tachycardia syndrome during graded tilt. Hypertension. 2015 Mar;65(3):636-43. doi: 10.1161/HYPERTENSIONAHA.114.04576. Epub 2014 Dec 15. PMID 25510829
- [Background] Anderson JW, Lambert EA, Sari CI, Dawood T, Esler MD, Vaddadi G, Lambert GW. Cognitive function, health-related quality of life, and symptoms of depression and anxiety sensitivity are impaired in patients with the postural orthostatic tachycardia syndrome (POTS). Front Physiol. 2014 Jun 25;5:230. doi: 10.3389/fphys.2014.00230. eCollection 2014. PMID 25009504
- [Background] Arnold AC, Haman K, Garland EM, Raj V, Dupont WD, Biaggioni I, Robertson D, Raj SR. Cognitive dysfunction in postural tachycardia syndrome. Clin Sci (Lond). 2015 Jan;128(1):39-45. doi: 10.1042/CS20140251. PMID 25001527
- [Background] Gibbons CH, Centi J, Vernino S, Freeman R. Autoimmune autonomic ganglionopathy with reversible cognitive impairment. Arch Neurol. 2012 Apr;69(4):461-6. doi: 10.1001/archneurol.2011.2372. Epub 2011 Dec 12. PMID 22158721
- [Background] Guaraldi P, Poda R, Calandra-Buonaura G, Solieri L, Sambati L, Gallassi R, Cortelli P. Cognitive function in peripheral autonomic disorders. PLoS One. 2014 Jan 17;9(1):e85020. doi: 10.1371/journal.pone.0085020. eCollection 2014. PMID 24465471
- [Result] Maier A, Schopen L, Thiel JC, Muller K, Fimm B, Schulz JB. Cognitive functioning in postural orthostatic tachycardia syndrome among different body positions: a prospective pilot study (POTSKog study). Clin Auton Res. 2023 Aug;33(4):459-468. doi: 10.1007/s10286-023-00950-0. Epub 2023 Jun 1. PMID 37261636